CLINICAL TRIAL: NCT01838226
Title: Randomized Controlled Trial of Group Prevention Coaching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CRE 12-285
Record Dates: First submitted 2013-04-18; First posted 2013-04-23 (Estimated); Results first posted 2020-05-19 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Cardiovascular Disease
Keywords: Chronic Disease; Prevention; cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases; Chronic Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group Prevention Clinics (Experimental): A group problem-solving intervention, with interval phone calls delivered to check in on goal progress and reinforce group learning. Groups will meet monthly for 6 months, and each patient will be called once between each group session. Each group will consist of 10 patients. Problem-solving teaches patients to overcome internal barriers to healthful behaviors. Problem solving will be combined, at all group sessions, with self-efficacy training, so that patients will be taught simultaneously to overcome both internal and external barriers. Participants will be asked to develop personal goals related to cardiovascular disease (CVD)-related behaviors (e.g., smoking and weight reduction).
  Interventions: Behavioral: Problem Solving
- Treatment as usual control (No Intervention): Usual VA care

INTERVENTIONS:
Behavioral: Problem Solving — A group problem-solving intervention, with interval phone calls delivered to check in on goal progress and reinforce group learning. Groups will meet monthly for 6 months, and each patient will be called once between each group session. Each group will consist of 10 patients. Problem-solving teaches patients to overcome internal barriers to healthful behaviors. Problem solving will be combined, at all group sessions, with self-efficacy training, so that patients will be taught simultaneously to overcome both internal and external barriers. Participants will be asked to develop personal goals related to CVD-related behaviors (e.g., smoking and weight reduction).
  Arms: Group Prevention Clinics

SUMMARY:
Prevention of cardiovascular disease is a primary focus of the Secretary's New Models of Care Transformational Initiative. However, prevention has been hard to accomplish. The VA is committed to using group visits to address a wide array of primary care problems. Coaching is a method to help Veterans set and reach health goals by helping them overcome barriers to behavior change. Coaching can be performed one-on-one or in groups. This study will test the effectiveness of a group prevention coaching (GPC) intervention in improving cardiovascular risk. GPCs will focus on changing a behavior of the patient's choice that is likely to lead to improvements in heart disease risk. The coach will adopt a problem-solving approach to helping Veterans make these improvements. The primary outcome will be change in 10-year risk of major cardiac event; the investigators will also assess improvements in food choice, physical activity and weight.

DETAILED DESCRIPTION:
Cardiovascular (CV) event prevention (e.g., myocardial infarction, cerebrovascular accident) remains the single most important public health problem in the United States, and cardiovascular disease is a leading cause of death among VA users. Improving the provision of prevention services is a primary focus of the Secretary's New Models of Care Transformational Initiative. However, prevention has been challenging to achieve. Multifactorial behavioral interventions are effective in treating a number of chronic illnesses (e.g., hypertension, diabetes), but less is known about their ability to reduce risk among patients without a unifying chronic illness. Group visits are an efficient, effective strategy for delivering a multifactorial behavior change intervention; the VA is committed to the group visit strategy to address a wide array of primary care problems. Groups have been shown to be an effective means of improving a number of outcomes in a number of individual diseases, but, again, their role in cardiovascular prevention among patients without a single common illness is unknown. Coaching is a type of multi-factorial behavioral intervention that involves goal-setting, and working to overcome barriers to behavior change. Coaching can be performed one-on-one, but coaching interventions have been delivered in group settings. The investigators have shown, in a 150-subject RCT, that group coaching plus individualized telephone coaching reduces cardiovascular risk, but the population in that study was very different from typical VA users. The investigators propose a three-site, two-arm randomized trial measuring the effectiveness of a group prevention coaching (GPC) intervention in improving cardiovascular risk, compared to VA usual care. The study will be performed at the Durham, Buffalo, and Syracuse VAMCs. Each arm will have 200 patients; patients will be VA users without prior history of cardiovascular event, but with at least 5% risk of such an event, and with either inadequately controlled hypertension or dyslipidemia, or current smoking. The GPC intervention will focus on changing a behavior of the patient's choice that is likely to lead to improvements in cholesterol, blood pressure, or to smoking cessation. Behaviors that will be reinforced will include but not be limited to healthy eating, decreased caloric intake, increased physical activity, stress reduction, and participatory decision making with physicians. Barriers to these behaviors will be identified. The coach will adopt a problem-solving approach to overcoming the above barriers and reinforcing the above behaviors; problem-solving is a well-described framework for behavior change. The GPC coach/interventionist for will be either the facility's Health Behavior Coordinator (HBC) or a person hired for the research enterprise but trained and credentialed identically to an HBC. All outcomes will be obtained at baseline, 6, and 12 months after enrollment by blinded research personnel. The primary outcome will be change in 10-year risk of fatal coronary event or non-fatal MI 6 months after enrollment, as measured by Framingham Risk Score. Key secondary outcomes will include dietary content by Food Frequency Questionnaire, physical activity as measured by International Physical Activity Questionnaire, and weight. The investigators will also determine if group cohesion, as measured by the Group Dynamics Inventory, influences the effectiveness of GPC. The investigators well also assess whether time spent in contact with a coach influences the effectiveness, by database log-in timekeeping strategies.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of inadequately controlled hypertension, as defined by an outpatient ICD-9 code of 401.x and a most recent blood pressure with either systolic > 140 mmHg or diastolic > 90 mmHg

  * OR (2) inadequately controlled dyslipidemia, as defined by most recent total cholesterol > 200 mg/dl or HDL cholesterol < 35 mg/dl
  * OR (3) current smoking, which can be identified using the CPRS Health Factor tied to the smoking clinical reminder.
* Medication-taking status for these illnesses is neither required nor excluded.

Exclusion Criteria:

* Subjects with very high risk of cardiovascular event, as determined by any personal history of coronary artery disease (CAD) or other major cardiovascular disease (ICD-9 code of 410-414, or 425-429)
* cerebrovascular disease (code 433-438)
* peripheral arterial disease (codes 440.x or 443.x)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Any
Enrollment: 401 (Actual)
Dates: Start 2014-08-29 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2019-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Edelman, MD MHS, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (2):
- United States (2):
  - VA Western New York Healthcare System, Buffalo, NY, Buffalo, New York
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
fully deidentified data will be shared as resources allow.

REFERENCES:
- [Result] Nieuwsma JA, Wray LO, Voils CI, Gierisch JM, Dundon M, Coffman CJ, Jackson GL, Merwin R, Vair C, Juntilla K, White-Clark C, Jeffreys AS, Harris A, Owings M, Marr J, Edelman D. A problem-solving intervention for cardiovascular disease risk reduction in veterans: Protocol for a randomized controlled trial. Contemp Clin Trials. 2017 Sep;60:42-50. doi: 10.1016/j.cct.2017.06.001. Epub 2017 Jun 23. PMID 28600161
- [Derived] Olsen MK, Stechuchak KM, Hung A, Oddone EZ, Damschroder LJ, Edelman D, Maciejewski ML. A data-driven examination of which patients follow trial protocol. Contemp Clin Trials Commun. 2020 Aug 13;19:100631. doi: 10.1016/j.conctc.2020.100631. eCollection 2020 Sep. PMID 32913914

RESULTS

PARTICIPANT FLOW:
Groups:
- Group Prevention Clinics: A group problem-solving intervention, with interval phone calls delivered to check in on goal progress and reinforce group learning. Groups will meet monthly for 6 months, and each patient will be called once between each group session. Problem-solving teaches patients to overcome internal barriers to healthful behaviors. Problem solving will be combined, at all group sessions, with self-efficacy training, so that patients will be taught simultaneously to overcome both internal and external barriers. Participants will be asked to develop personal goals related to cardiovascular disease (CVD)-related behaviors (e.g., smoking and weight reduction). Problem-solving teaches patients to overcome internal barriers to healthful behaviors. Problem solving will be combined, at all group sessions, with self-efficacy training. Participants will be asked to develop personal goals related to CVD-related behaviors (e.g., smoking and weight reduction).
Period: Overall Study
Arm/Group | Group Prevention Clinics | Treatment as Usual Control
Started | 202 | 199
Completed | 126 | 128
Not Completed | 76 | 71

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group Prevention Clinics | Treatment as Usual Control | Total
Number analyzed (Participants) | 202 | 199 | 401
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (11.1) | 61.9 (9.2) | 62.4 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 19 | 40
  Male | 181 | 180 | 361
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 4 | 11
  Not Hispanic or Latino | 195 | 195 | 390
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 60 | 69 | 129
  White | 130 | 116 | 246
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 12 | 14 | 26
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 202 | 199 | 401
Framingham Risk Score [Mean (Standard Deviation); unit: percent risk of event] — These are baseline Framingham Risk Score data. Scores range from 0 - 100, as this is a percentage of risk. Higher scores are worse, as they represent higher risk.
  percent risk of event | 28.9 (15.2) | 29.5 (17.2) | 29.2 (16.2)

OUTCOME MEASURES:

1. Primary Outcome: Risk of Fatal Coronary Event or Non-fatal MI
Description: The primary outcome will be 10-year risk of fatal coronary event or non-fatal MI 6 months after enrollment, as measured by Framingham Risk Score. Scores range from 0 - 100, as this is a percentage of risk. Higher scores are worse, as they represent higher risk.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percent risk of major cv event in 10 yrs
Arm/Group | Group Prevention Clinics | Treatment as Usual Control
Number analyzed (Participants) | 202 | 199
percent risk of major cv event in 10 yrs | 27.0 (17.2) | 26.3 (15.5)
Statistical Analysis 1: Comparison: Group Prevention Clinics vs Treatment as Usual Control; Test type: Superiority; p = 0.50, Mixed Models Analysis; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-1.3 to 2.8]

2. Secondary Outcome: Patient Activation Measure
Description: Measure of self-efficacy. Scored from 0-100, with 100 being higher self-efficacy and a better outcome.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group Prevention Clinics | Treatment as Usual Control
Number analyzed (Participants) | 202 | 199
units on a scale | 62.1 (11.5) | 62.6 (12.2)
Statistical Analysis 1: Comparison: Group Prevention Clinics vs Treatment as Usual Control; Test type: Superiority; Mixed Models Analysis; Mean Difference (Net) = 0.9, 95% CI 2-sided [-1.3 to 3.1]

3. Secondary Outcome: Risk of Fatal Coronary Event or Non-fatal MI
Description: The primary outcome will be 10-year risk of fatal coronary event or non-fatal MI 12 months after enrollment, as measured by Framingham Risk Score. Scores range from 0 - 100, as this is a percentage of risk. Higher scores are worse, as they represent higher risk.
Time Frame: 12 month
Measure: Mean (Standard Deviation); unit: percent risk of cv event in 10 years
Arm/Group | Group Prevention Clinics | Treatment as Usual Control
Number analyzed (Participants) | 202 | 199
percent risk of cv event in 10 years | 25.7 (15.4) | 28.2 (16.8)
Statistical Analysis 1: Comparison: Group Prevention Clinics vs Treatment as Usual Control; Test type: Superiority; Mean Difference (Net) = -2.6, 95% CI 2-sided [-4.9 to -0.2]

ADVERSE EVENTS:
Time Frame: 12 months
Description: Adverse events were assessed without regard to specific adverse event terms.
Arm/Group | Group Prevention Clinics | Treatment as Usual Control
All-Cause Mortality (participants affected / at risk) | 1/202 | 0/199
Serious Adverse Events (participants affected / at risk) | 1/202 | 0/199
Other Adverse Events (participants affected / at risk) | 0/202 | 0/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group Prevention Clinics (N=202) | Treatment as Usual Control (N=199)
death (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-26): https://cdn.clinicaltrials.gov/large-docs/26/NCT01838226/Prot_SAP_000.pdf